CLINICAL TRIAL: NCT00671359
Title: An Open-Label, Single-Dose, Two-Treatment, Randomized, Two-Way Crossover, Safety, Tolerance, and Pharmacokinetic Study of TR-701 in Normal Healthy Adults in the Fed and Fasted State
Brief Title: Food Effects of Single Oral Dose of 600mg TR-701
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1986-023; TR701-103 (Other: TriusRX Unique ID)
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Healthy
Keywords: Food effects
MeSH Terms: interventions — tedizolid phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- after fast (Experimental): Administration of a single oral dose of 600mg TR-701 to subjects in the fasted state.
  Interventions: Drug: TR-701 600mg
- After high fat food (Experimental): Administration of a single oral dose of 600mg TR-701 to subjects in the fed state.
  Interventions: Drug: TR-701 600mg

INTERVENTIONS:
Drug: TR-701 600mg — TR-701 600mg

SUMMARY:
This is an evaluation of the safety, tolerance, and pharmacokinetics of single oral doses of TR-701 given to normal, healthy, adult volunteers in the fed and fasted state.

DETAILED DESCRIPTION:
Subjects will receive the following treatments in a crossover design:

Treatment A: Three 200-mg capsules (600-mg dose) of TR-701 administered orally with 240 mL room temperature tap water after at least a 10-hour fast.

Treatment B: Three 200-mg capsules (600-mg dose) of TR-701 administered orally with 240 mL room temperature tap water following a high-fat meal preceded by at least a 10-hour fast.

Descriptive statistics will be calculated for PK parameters where available, including Cmax, Tmax, AUC0-t, and AUC0-inf. Minimum, maximum, mean, and median values will be determined and standard deviations will be calculated. Where data are available, food effect will be examined between test (fed state) and reference (fasted state) groups.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 20 to 29.9 kg/m2
* Females must be either postmenopausal for at least 1 year, surgically sterile for at least 90 days, or agree to use an acceptable method of birth control

Exclusion Criteria:

* history or clinical manifestations of any clinically significant medical disorder
* history of hypersensitivity or allergies to any drug compound
* history of stomach or intestinal surgery or resection
* history of alcoholism or drug addiction within 1 year
* pregnancy, lactation, or breastfeeding
* use of any tobacco-containing or nicotine-containing products within 6 months
* use of any other medications
* use of alcohol-containing, grapefruit-containing, or caffeine-containing foods or beverages; or foods or beverages with high levels of tyramine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-03-10 (Actual); Primary Completion 2008-05-15 (Actual); Study Completion 2008-05-15 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of TR-701 600mg given as a single oral dose. | 4 days

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of single doses of TR-701 and its microbiologically active moiety, TR-700, in healthy adult volunteers in the fed and fasted state | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Berry, MD, Principal Investigator — Covance CRU
Locations (1):
- Covance CRU, San Diego, California, United States

REFERENCES:
- [Derived] Flanagan SD, Bien PA, Munoz KA, Minassian SL, Prokocimer PG. Pharmacokinetics of tedizolid following oral administration: single and multiple dose, effect of food, and comparison of two solid forms of the prodrug. Pharmacotherapy. 2014 Mar;34(3):240-50. doi: 10.1002/phar.1337. Epub 2013 Aug 7. PMID 23926058